CLINICAL TRIAL: NCT05905796
Title: Low-cost Detection of Dementia Using Electronic Health Records Data: Validation and Testing of the Electronic Health Record Risk of Alzheimer's and Dementia Assessment Rule (eRADAR) Algorithm in a Pragmatic, Patient-centered Trial.
Brief Title: The Brain Health Study: A Pragmatic, Patient-Centered Trial
Acronym: eRADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R01AG069734 (NIH); 1R01AG069734 (NIH)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health Intervention (Experimental): Calculate eRADAR scores using EHR data to identify eligible individuals Invite eligible individuals for brain health assessment visit Enter results of brain health assessment visit into EHR Provide summary of results and recommended next steps to the Primary Care Physician and participant
  Interventions: Other: Brain Health Assessment
- Usual Care (No Intervention): Usual care Individuals who meet eligibility criteria will receive usual care.

INTERVENTIONS:
Other: Brain Health Assessment — Research interventionists, who will be trained and licensed health practitioners (e.g., social workers), will ask participants about changes in memory or thinking and daily function, screen for depression, and administer a standard cognitive screening test. Research interventionalists will use a standardized note template to document results in the participant's EHR. Research interventionists will notify participants and PCPs if follow-up is recommended.
  Arms: Brain Health Intervention

SUMMARY:
The eRADAR Brain Health Study seeks to refine and test a novel, low-cost strategy for increasing dementia detection within primary care.

DETAILED DESCRIPTION:
Detailed description: eRADAR stands for "electronic health record (EHR) Risk of Alzheimer's and Dementia Assessment Rule." It is a low-cost tool or algorithm that uses readily available EHR data elements to identify high-risk patients. The investigators will conduct a pragmatic randomized controlled trial to assess the impact of implementing eRADAR as part of a supported outreach process on dementia detection rates. The investigators will also explore the impact of eRADAR implementation on healthcare utilization and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* No prior diagnosis of dementia (defined from EHR diagnosis codes) and not receiving medications for dementia
* Active patient at participating clinic
* Adequate data to calculate eRADAR score

Exclusion Criteria:

- Currently receiving hospice care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1271 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
New dementia diagnosis | 12 months after index date
  Rate of new dementia diagnosis identified from the electronic health record (EHR) using prespecified set of ICD-10 codes

SECONDARY OUTCOMES:
Number of primary care visits | 6 months after index date
  Defined from EHR data
Number of dementia-related laboratory tests performed | 6 months after index date
  Defined from EHR data
Number of dementia-related neuroimaging tests performed | 6 months after index date
  Defined from EHR data
Number of specialty visits or referrals for dementia assessment | 6 months after index date
  Defined from EHR data
Percent of participants who receive new medications for dementia | 6 months after index date
  Defined from medication orders or dispensings in the electronic health record
Number of urgent care and emergency department visits | 1 year after index date
  Defined from EHR data
Number of inpatient days | 1 year after index date
  Defined from EHR data
Number of scheduled visits missed | 1 year after index date
  Clinic "no shows"
Proportion of days covered for current prescriptions | 1 year after index date
  Standard measure of medication adherence
New dementia diagnosis (secondary definitions) | 6 months after index date
  Rate of new dementia diagnosis identified from the electronic health record (EHR) using prespecified set of ICD-10 codes
New dementia diagnosis (secondary definitions) | 18 months after index date
  Rate of new dementia diagnosis identified from the electronic health record (EHR) using prespecified set of ICD-10 codes
New diagnosis of mild cognitive impairment | 12 months after index date
  Rate of new diagnosis of mild cognitive impairment following the intervention, defined from EHR data
Proportion of people offered a brain health visit who accept and attend the visit | 3 months after invitation mailed
  Rate of accepting brain health visit
Positive predictive value of eRADAR algorithm | 12 months after index date
  Proportion of people with a high risk eRADAR Score who attend a brain health visit who are diagnosed with dementia

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Barnes, PhD, Principal Investigator — University of California, San Francisco; Sascha Dublin, MD, PhD, Principal Investigator — KP Washington Health Research Institute
Locations (3):
- United States (3):
  - UCSF Primary Care at China Basin, San Francisco, California
  - Division of General Internal Medicine, San Francisco, California
  - Women's Health Primary Care, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Plan description: This Individual Participant Data (IPD) plan applies to all quantitative study data, such as data collected specifically for the study and those derived from electronic health records (EHR), as well as the data collected via planned study surveys, which include only short qualitative free-text fields. The investigators do not plan to share transcripts from in-depth qualitative interviews or recorded study assessment visits.
  Data will be maintained on secure servers behind the firewalls at the two study sites: Kaiser Permanente Washington (KPWA) and the University of California, San Francisco (UCSF). De-identified or limited datasets containing individual-level data on which publications are based will be made available to qualified researchers for specified analyses. The investigators will make the data available to users only under a data-use agreement (DUA).
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested after the primary study paper is accepted for publication, up until 5 years after study completion.
Access Criteria: Individuals interested in using KPWA data will be required to complete a standard form, sign a Data Use Agreement (DUA) and provide documentation of IRB approval. Data may then be accessed by qualified researchers via KPWA's Secure File Transfer (SFT) site. User registration will be required in order to access or download data files. As part of the registration process, users must agree to the conditions of use governing access to the data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgment of the data resource.
  Individuals interested in using UCSF data will be required to complete the same data request form. The UCSF Industry Contracts Division (ICD), which oversees incoming and outgoing transfer of all UCSF data, will review the form for compliance with UCSF policies.

REFERENCES:
- [Background] Dublin S, Greenwood-Hickman MA, Karliner L, Hsu C, Coley RY, Colemon L, Carrasco A, King D, Grace A, Lee SJ, Walsh JME, Barrett T, Broussard J, Singh U, Idu A, Yaffe K, Boustani M, Barnes DE. The electronic health record Risk of Alzheimer's and Dementia Assessment Rule (eRADAR) Brain Health Trial: Protocol for an embedded, pragmatic clinical trial of a low-cost dementia detection algorithm. Contemp Clin Trials. 2023 Dec;135:107356. doi: 10.1016/j.cct.2023.107356. Epub 2023 Oct 17. PMID 37858616
- [Background] Lee SJ, Larson EB, Dublin S, Walker R, Marcum Z, Barnes D. A Cohort Study of Healthcare Utilization in Older Adults with Undiagnosed Dementia. J Gen Intern Med. 2018 Jan;33(1):13-15. doi: 10.1007/s11606-017-4162-3. No abstract available. PMID 28849435
- [Background] Barnes DE, Zhou J, Walker RL, Larson EB, Lee SJ, Boscardin WJ, Marcum ZA, Dublin S. Development and Validation of eRADAR: A Tool Using EHR Data to Detect Unrecognized Dementia. J Am Geriatr Soc. 2020 Jan;68(1):103-111. doi: 10.1111/jgs.16182. Epub 2019 Oct 14. PMID 31612463
- [Background] Coley RY, Smith JJ, Karliner L, Idu AE, Lee SJ, Fuller S, Lam R, Barnes DE, Dublin S. External Validation of the eRADAR Risk Score for Detecting Undiagnosed Dementia in Two Real-World Healthcare Systems. J Gen Intern Med. 2023 Feb;38(2):351-360. doi: 10.1007/s11606-022-07736-6. Epub 2022 Jul 29. PMID 35906516